CLINICAL TRIAL: NCT00593567
Title: A Study to Investigate the Safety and Efficacy of a Topical Gentamicin-Collagen Sponge Compared to Levofloxacin in Diabetic Patients With a Mild Infection of a Lower Extremity Skin Ulcer
Brief Title: Safety and Efficacy of an Antibiotic Sponge in Diabetic Patients With a Mild Infection of a Foot Ulcer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INN-TOP-001
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Daily topical gentamicin sponge and standard daily wound care
  Interventions: Drug: gentamicin-collagen sponge
- B (Active Comparator): Daily oral levofloxacin 750 mg and standard daily wound care
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: gentamicin-collagen sponge — Inserted daily into open ulcer
  Arms: A
Drug: Levofloxacin — 750mg oral levofloxacin daily
  Arms: B

SUMMARY:
The purpose of this study is to determine whether the gentamicin-collagen sponge when combined with standard of daily wound care is safe and effective in treating mildly infected skin ulcers compared to treatment with an oral antibiotic (levofloxacin) and standard daily wound care.

DETAILED DESCRIPTION:
Infected skin ulcers in patients with diabetes can be very debilitating because they are difficult to heal. Diabetic ulcers are responsible for frequent health care visits, and are a major predictor of amputation. Diabetic ulcers can be caused by a patient's inability to sense pain or warmth as well as peripheral vascular disease, which causes diminished blood flow to the foot. Early aggressive treatment is necessary to treat infection and prevent the need for amputation.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin-collagen sponge is a thin flat sponge made out of collagen that comes from cow tendons and containing gentamicin. When applied to an open ulcer, the collagen breaks down and the gentamicin is released into the ulcer, but very little is absorbed into the blood stream. The high levels of gentamicin in the open infected ulcer may help treat the infection.

In this study, all subjects will be given the necessary supplies and taught how to take care of their foot ulcer. Subjects who are randomly assigned to the gentamicin-collagen sponge treatment group will place a gentamicin-collagen sponge on their ulcer during daily wound care. Subjects who are randomly assigned to the oral levofloxacin treatment group will also perform daily wound care, but they will not be given the gentamicin-collagen sponge. Instead they will be given the antibiotic, levofloxacin to take by mouth during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Is a man or woman aged 18 to 80 years.
* Has diabetes mellitus, according to the American Diabetes Association criteria.
* Has a single infected skin ulcer below the knee, defined as "mild" by the Infectious Disease Society of America (IDSA) Guidelines, for whom, in the Investigator's judgment, topical or oral antimicrobial therapy is appropriate (Mild infection severity: The presence of ≥ 2 manifestations of inflammation (purulence or erythema, pain, tenderness, warmth or induration) but any cellulitis/erythema extends ≤ 2 cm around the ulcer, and the infection is limited to the skin or superficial subcutaneous tissue, with no other local complications or acute, systemic illness).
* Has had an x-ray of the infected area within the 2 days immediately preceding or at Visit 1 (Baseline/Randomization) that is negative for osteomyelitis.
* Meets the certain minimal laboratory criteria
* Has an ankle-brachial index (ABI) ≥ 0.7 and ≤ 1.3. (Note: Patients with ABI < 0.7 or > 1.3 may be included if they have either a transcutaneous oxygen pressure or a toe pressure ≥ 40 mm Hg on the limb with the target ulcer.)
* If female, is nonpregnant (negative pregnancy tests at the Baseline/Randomization Visit) and nonlactating.
* If female, is either not of childbearing potential (defined as postmenopausal for ≥ 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing 1 of the following medically-acceptable methods of birth control and agrees to continue with the regimen throughout the duration of the study:

  * Oral, implantable or injectable contraceptives for 3 consecutive months before the Baseline/Randomization Visit
  * Total abstinence from sexual intercourse (≥ 1 complete menstrual cycle before the Baseline/Randomization Visit)
  * Intrauterine device (IUD)
  * Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* Willing to return to the study facility for the Final Study Visit.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study

Exclusion Criteria:

* Has a known history of hypersensitivity to gentamicin (or other systemic aminoglycosides) or levofloxacin or drugs in the same class, or any of the test article or reference product components.
* Has a known hypersensitivity to bovine collagen.
* Has any uncontrolled illnesses that, in the opinion of the Investigator, would interfere with interpreting the results of the study.
* Has an infecting pathogen known to be intermediate or resistant in vitro to levofloxacin. Patients enrolled into the study presumptively will be discontinued if their cultured organism is intermediate or resistant to levofloxacin.
* Has a target ulcer with a wound size > 5 × 5 cm.
* Has gangrenous tissue of the affected limb that cannot be removed with a single debridement.
* Has a wound associated with prosthetic material or device.
* Received any topical or systemic antimicrobial therapy within the 2 weeks prior to study entry (Visit 1 [Day 1]).
* Has documented osteomyelitis.
* If severely immunocompromised, may be excluded at the discretion of the Investigator.
* Has a history of alcohol or substance abuse in the past 12 months.
* Is undergoing dialysis (renal or peritoneal) or has history of kidney transplant.
* Has a history of myasthenia gravis or other neurological condition where gentamicin use is contraindicated as determined by the Investigator.
* Has a history of epilepsy
* Has a history of tendon disorders related to fluoroquinolone administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Chesapeake Research Group LLC, Pasadena, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gentamicin Sponge: Daily topical gentamicin sponge and standard daily wound care
  gentamicin-collagen sponge: Inserted daily into open ulcer
- Levofloxacin: Daily oral levofloxacin 750 mg and standard daily wound care
  Levofloxacin: 750mg oral levofloxacin daily
Period: Overall Study
Arm/Group | Gentamicin Sponge | Levofloxacin
Started | 48 | 22
Completed | 28 | 12
Not Completed | 20 | 10
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 13 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gentamicin Sponge | Levofloxacin | Total
Number analyzed (Participants) | 47 | 22 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (10.54) | 58.9 (14.04) | 59.4 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 12 | 41
  Male | 18 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 40 | 17 | 57
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Outcome of "Clinical Cure"
Description: Number of Participants with a clinical outcome of "clinical cure" at final visit. Clinical Cure is defined as positive clinical response and with pathogen eradication.
Time Frame: Final Study Visit (Day 21 [or 28 or 35])
Population: Modified Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 34 | 15
Participants | 14 | 7

2. Secondary Outcome: Number of Participants With a Clinical Outcome of "Clinical Cure" in Each Treatment Group
Description: Number of participants with a clinical outcome of "clinical cure" in each treatment group at/by each time point (except the Final Study Visit). Clinical Cure is defined as positive clinical response and with pathogen eradication.
Time Frame: Each time point (Day 3, 7 [14 and 21 if necessary])
Population: Modified intent to treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 34 | 15
Participants
  Visit 2 Day 3 | 0 | 0
  Visit 3 Day 7 | 4 | 0
  Visit 4 Day 14 | 4 | 6
  Visit 5 Day 21 | 8 | 0
  Final Study Visit | 14 | 7

3. Secondary Outcome: Time to Baseline Pathogen Eradication
Time Frame: assessed at each time point on days 7, 14, 21, time to pathogen eradication from baseline up to day 21 reported
Population: mITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 31 | 14
Days | 7.0 [7.0 to 8.0] | 14.5 [7.0 to NA] — Upper boundary not reached

4. Secondary Outcome: Number of Participants With Complete Wound Closure by Each Visit
Time Frame: At each timepoint Day 3, 7, 14 & 21
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 34 | 15
Participants
  Visit 2 Day 3 | 0 | 0
  Visit 3 Day 7 | 2 | 0
  Visit 4 Day 14 | 3 | 2
  Visit 5 Day 21 | 4 | 2

5. Secondary Outcome: Time to Clinical Cure
Description: Time to Clinical Cure is measured by days to the first observed cure. Clinical Cure is defined as positive clinical response and with pathogen eradication.
Time Frame: Actual time assessed (Day 1, 3, 7 [14 and 21 if necessary] and Day 21 [or 28 or 35])
Population: Modified ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 34 | 15
Days | 22.0 [21.0 to NA] — 17 patients censored | NA [14.0 to NA] — 8 out of 15 patients censored

6. Secondary Outcome: Time to Pathogen Eradication
Description: Time to Baseline Pathogen Eradication summed
Time Frame: Actual time assessed (Day 1-21
Population: Micro Modified Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 30 | 14
Days | 7.0 [7.0 to 8.0] | 14.5 [7.0 to NA] — not able to calculate high boundary

7. Secondary Outcome: Time to Positive Clinical Response
Time Frame: (Day 1, 3, 7 [14 and 21 if necessary] and Day 21 [or 28 or 35])
Population: mITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gentamicin Sponge | Levofloxacin
Number analyzed (Participants) | 34 | 15
Days | 2.0 [2.00 to 3.0] | 3.0 [2.0 to 3.0]

ADVERSE EVENTS:
Time Frame: about 35 days.
Arm/Group | Gentamicin Sponge | Levofloxacin
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/22
Other Adverse Events (participants affected / at risk) | 15/47 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gentamicin Sponge (N=47) | Levofloxacin (N=22)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Odema peripheral (General disorders) | 0 (0) | 1 (1)
Pitting oedema (General disorders) | 0 (0) | 1 (1)
Naspoharygitis (Infections and infestations) | 1 (1) | 2 (2)
Bacterial infections (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract infections (Infections and infestations) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriatiosn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin lacerations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Would complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Red blood cell urine positive (Investigations) | 0 (0) | 1 (1)
white blood cell count decreased (Investigations) | 1 (1) | 0 (0)
white blood cells urine positive (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No